CLINICAL TRIAL: NCT00897637
Title: Categorization of Wilms Tumors by Genetic Expression
Brief Title: Gene Expression Profiles to Categorize Wilms Tumors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN03B1; NCI-2009-00415 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000349184 (Other: Clinical Trials.gov); COG-AREN03B1 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Stage I Wilms Tumor; Stage II Wilms Tumor; Stage III Wilms Tumor; Stage IV Wilms Tumor; Stage V Wilms Tumor
MeSH Terms: conditions — Wilms Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Three hundred tumor specimens are analyzed for genetic expression profiles using Affymetrix assays. Specific genes are identified as classifiers and analyzed using tissue arrays. An additional 300 specimens are examined for gene expression and categorized according to the classifiers.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This laboratory study is using gene expression profiling to identify different categories of Wilms tumors. Studying the genes expressed in samples of tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Identify new molecular categories of Wilms tumor (WT) based on the gene expression profiles of samples from patients with this disease.

II. Develop a classifying system (classifier) that will predict a defined number of clinically relevant categories based on expression of an established set of genes.

III. Confirm and test the classifier with further analysis of the genes by several different methodologies, using additional patient samples that are outside of the case/cohort but which possess the clinically or scientifically relevant parameter.

IV. Validate the use of the classifier to predict defined groups within a second set of samples (for which investigators are blinded to the clinical and biological data) by subsequent comparison with true incidence of pertinent markers.

OUTLINE:

Three hundred tumor specimens are analyzed for genetic expression profiles using Affymetrix assays. Specific genes are identified as classifiers and analyzed using tissue arrays. An additional 300 specimens are examined for gene expression and categorized according to the classifiers.

ELIGIBILITY:
Inclusion Criteria:

* Specimens from patients previously enrolled as "On Study" or "Followed Biology Only" on protocol NWTSG-5 (COG-Q9401)

  * Study follow-up data for disease status available
* National Wilms Tumor Study Group/Children's Oncology Group pathology review showing "favorable" histology
* Sufficient biology samples available without using biology bank reserves

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Specimens from patients previously enrolled as "On Study" or "Followed Biology Only" on protocol NWTSG-5 (COG-Q9401)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2004-02; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
New molecular categories of Wilms tumor identified and measured by gene expression profiles | Up to 6 years
Identification of genes that as a whole provide strong prediction of outcomes of interest | Up to 6 years
  Supervised methods such as CART or Shrunken Centroid Classifier will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Perlman, MD, Principal Investigator — Children's Oncology Group
Locations (2):
- United States (2):
  - Children's Oncology Group, Arcadia, California
  - Saint Mary's Hospital, West Palm Beach, Florida